CLINICAL TRIAL: NCT01950988
Title: Effectiveness and Satisfaction-adaptability of a Novel Concept for a Manual Toothbrush Broscyl®: Randomised Clinical Trial in Children, Adults and Elderly People
Brief Title: Effectiveness of a Novel Concept for a Manual Toothbrush Broscyl®
Acronym: BROSCYL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ZWETYENGA PHRC IR 2011
Record Dates: First submitted 2013-08-27; First posted 2013-09-26 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Children (Other)
  Interventions: Device: Manual toothbrush reference; Procedure: Measure of the dental plaque; Device: Manual toothbrush Broscyl®
- Adults (Other)
  Interventions: Device: Manual toothbrush reference; Procedure: Measure of the dental plaque; Device: Manual toothbrush Broscyl®
- Elderly people (Other)
  Interventions: Device: Manual toothbrush reference; Procedure: Measure of the dental plaque; Device: Manual toothbrush Broscyl®

INTERVENTIONS:
Device: Manual toothbrush reference
Procedure: Measure of the dental plaque
Device: Manual toothbrush Broscyl®

SUMMARY:
The aim is to determine the efficacy and the satisfaction/adaptability of the manual Broscyl® toothbrush as compared with a standard " soft " manual toothbrush ADA (American Dental Association) reference using the modified Stillman brushing technique, in children, adults and elderly persons, after 3 months of daily use.

ELIGIBILITY:
Inclusion Criteria:

* Children attending school aged between 8 and 15 years
* OR adults aged from 18 to 45 years
* OR elderly persons aged more than 65 years old
* Presenting at least one incisive, one canine, one premolar and one molar in each quadrant
* Able to brush their own teeth at least twice a day
* Persons who have provided written informed consent
* Persons covered by the national health insurance agency

Exclusion Criteria:

* Persons with acute periodontal disease
* Persons in a period of postsurgical healing
* Persons with an acute oral pain syndrome
* Persons undergoing orthodontic treatment with a fixed brace
* Persons not covered by the national health insurance agency
* Pregnant women
* The use of adjuvants

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2013-07-16 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2016-06-08 (Actual)

PRIMARY OUTCOMES:
Measurement of the dental plaque index | up to 3 months

SECONDARY OUTCOMES:
Patient satisfaction | up to 3 months
  self-completed questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France